CLINICAL TRIAL: NCT05405855
Title: eLIFEwithIBD (Living With Intention, Fullness and Engagement With Inflammatory Bowel Disease): The Impact of an ICT-based Intervention on Physical and Mental Health
Brief Title: eLIFEwithIBD - Living With Intention, Fullness and Engagement With Inflammatory Bowel Disease (Online)
Acronym: eLIFEwithIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Inês A Trindade, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINEICC-2-IAT
Record Dates: First submitted 2022-05-27; First posted 2022-06-06 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The eLIFEwithIBD intervention is an ACT, mindfulness and compassion eHealth intervention for people with inflammatory bowel disease (IBD). The eLIFEwithIBD intervention is delivered through 9 sessions available on an online platform throughout a 9-week period. Each session is composed of real-image videos, texts with illustrative images, exercises in editable text format, and audio files with the experiential exercises and practices targeting topics such as acceptance, mindfulness, compassion, and gratitude.
  Participants in this group also continue to receive a standard, personalised treatment for IBD.
  Interventions: Behavioral: eLIFEwithIBD
- Control Group (No Intervention): Treatment as Usual (TAU) - Standard, personalised treatment for inflammatory bowel disease.

INTERVENTIONS:
Behavioral: eLIFEwithIBD — eLIFEwithIBD program is a psychotherapeutic programme based on Acceptance, Mindfulness and Compassion for inflammatory bowel disease patients.
  Arms: Experimental Group

SUMMARY:
This study aims to test the acceptability and preliminary efficacy of an online intervention (eLIFEwithIBD) developed for people with inflammatory bowel disease (IBD). The eLIFEwithIBD intervention is an adaptation of the LIFEwithIBD program (delivered in an in-person group format; Trindade et al., 2021), being an ACT, mindfulness, and compassion-based intervention. The eLIFEwithIBD intervention comprises nine sessions focusing on education about IBD, the functioning of the mind, emotions, and fatigue; acceptance of internal experiences; willingness; emotion regulation; values clarification; committed action; mindfulness; compassion; and gratitude. These topics are addressed through videos with therapists, texts, and experiential exercises.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65;
* IBD diagnosis (at least from 6 months prior);
* regular access to a computer with internet;
* able to write and read in Portuguese, and give informed consent.

Exclusion Criteria:

* diagnosis of a psychiatric disorder (major depressive disorder, psychotic disorder, bipolar disorder, substance abuse), or suicidal ideation (assessed by the Patient Health Questionnaire-9);
* current psychotherapy use;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Psychological distress (DASS-21; Lovibond & Lovibond, 1995) | From Baseline to 4-months follow-up
  The DASS-21 is a 21-item measure of depressive (e.g., "I felt I wasn't worth much as a person"), anxiety (e.g., "I felt scared without any good reason"), and stress (e.g., "I found it hard to wind down") symptoms during the precedent week, using a 4-point scale [ranging from "did not apply to me at all" (0) to "applied to me very much, or most of the time" (3)].

SECONDARY OUTCOMES:
Perception of Quality of Life - EUROHIS-QOL 8-item index (Power, 2017); Inflammatory Bowel Disease Questionnaire - UK version (IBDQ-UK; Cheung et al., 2000) | From Baseline to 4-months follow-up
  The EUROHIS-QOL 8-item index is a quality of life measure composed of eight items (regarding general health, energy, daily living activity, overall quality of life, finances, social relationships, self-esteem, and home) which were extracted from the WHOQOL-Bref. Each item has an individualized 5-point Likert scale (the same response scales used in the WHOQOL-bref).
  The Inflammatory Bowel Disease Questionnaire-UK version (IBDQ-UK), which is the Anglicized 30-item version of the IBDQ (79, 80), an IBD-specific quality of life instrument. Each item is rated on a 4-point scale (three questions have an additional "non-applicable" option available) ranging from "no, no at all/none" (0) to "on 8 to 14 days (i.e., more than every other day)/Yes, all of the time" (4). Participants are asked to answer questions regarding their IBD and how it has affected their lives during the previous 2 weeks.
Chronic illness-related shame (Chronic Illness-related Shame Scale - CISS, Trindade et al., 2017) | From Baseline to 4-months follow-up
  The CISS is a 7-item unidimensional scale that was specifically designed to evaluate shame associated with the experience of having a chronic illness and/or its related symptoms (e.g., "I feel inadequate because of my illness and symptoms," "I'm ashamed of talking with others about my illness or symptoms," "I feel that my illness is embarrassing"). Each item is rated on a 5-point Likert scale [from"Never true" (0) to "Always true" (4)].
IBD symptom perception (IBD symptoms scale, Trindade et al., 2019) | From Baseline to 4-months follow-up
  IBD symptoms scale is a 16-item self-report Portuguese scale which was developed to evaluate the frequency of IBD symptoms during the precedent month (e.g., fatigue, abdominal pain and bloating, flatulence, diarrhea, nausea or vomiting, fever, the urgency to evacuate). Each item is rated on a 7-point scale [ranging from "Never" (0) to "Always" (6)].
Functional impairment (Work and Social Adjustment Scale - WSAS; Mundt et al., 2002) | From Baseline to 4-months follow-up
  The Work and Social Adjustment Scale (WSAS) is a 5-item measure of perceived functional impairment in daily activities, such as work, family, interpersonal relations, social and private leisure activities, and home management. Each item is rated on a 9-point scale ["Not at all" (0) to "Very severely" (8)].

OTHER OUTCOMES:
Usability - System Usability Scale (SUS; Brooke, 1986) | 9 weeks
  SUS is a 10-item self-report scale aimed to evaluate product and user interface usability (e.g., the confidence and ease of use of the plafaform). Items are rated on a 5-point scale ranging from completely disagree (1) to completely agree (5).
Acceptability and Feasibility - The Acceptability and Feasibility Measures (Weiner et al., 2017) | 9 weeks
  A four-item self-report instrument measures the acceptability and feasibility of the intervention. Items are answered using a 5-point Likert scale ranging from completely disagree (1) to completely agree (5).

CONTACTS AND LOCATIONS:
Locations (1):
- Inês Trindade, Coimbra, Portugal

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Ferreira C, Pereira J, Matos-Pina I, Skvarc D, Galhardo A, Ferreira N, Carvalho SA, Lucena-Santos P, Rocha BS, Oliveira S, Portela F, Trindade IA. eLIFEwithIBD: study protocol for a randomized controlled trial of an online acceptance and commitment therapy and compassion-based intervention in inflammatory bowel disease. Front Psychol. 2024 Aug 9;15:1369577. doi: 10.3389/fpsyg.2024.1369577. eCollection 2024. PMID 39184944